CLINICAL TRIAL: NCT05999006
Title: A Prospective, Multicenter, Clinical Trial Designed to Evaluate the Safety and Feasibility of the ELIOS System to Reduce Intraocular Pressure in Patients With Primary Open-Angle Glaucoma as a Standalone Procedure
Brief Title: Safety and Feasibility of the ELIOS System in POAG Patients
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Elios Vision, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: EP-02
Record Dates: First submitted 2023-08-11; First posted 2023-08-21 (Actual); Last update posted 2025-06-17 (Actual); Status verified 2025-06

CONDITIONS: Glaucoma, Primary Open Angle
MeSH Terms: conditions — Glaucoma, Open-Angle

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes

ARMS (1):
- ELIOS Procedure (Experimental): ELIOS Procedure
  Interventions: Device: ELIOS Procedure

INTERVENTIONS:
Device: ELIOS Procedure — Treatment with the ELIOS System

SUMMARY:
Evaluation of the safety and effectiveness of the ELIOS System procedure to reduce intraocular pressure (IOP) in adult subjects with mild to moderate primary open-angle glaucoma (POAG)

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of mild to moderate POAG
* Medicated IOP of <=24 mmHg
* Shaffer angle grade of III or IV
* CD ratio <=0.8
* At least 45 years old

Exclusion Criteria:

* Closed-angle and secondary glaucomas
* Prior incisional glaucoma surgery, intraocular surgery, or corneal surgery
* Cannot undergo medication washout in the study eye
* Diagnosis of degenerative visual disorders Non-study eye with BCVA worse than 20/80 Known corticosteroid responder Pregnant or nursing women; or women of childbearing potential not using medically acceptable birth control

Min Age: 45 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 65 (Estimated)
Dates: Start 2023-10-18 (Actual); Primary Completion 2026-04 (Estimated); Study Completion 2026-04 (Estimated)

PRIMARY OUTCOMES:
Proportion of subjects who achieve a decrease in mean diurnal IOP (DIOP) from baseline of at least 20% on the same or fewer medications | 12 Months
  Proportion of subjects who achieve a decrease in mean diurnal IOP (DIOP) from baseline of at least 20% on the same or fewer medications
Mean Change in DIOP from baseline on the same or fewer medications | 12 Months
  Mean Change in DIOP from baseline on the same or fewer medications

CONTACTS AND LOCATIONS:
Overall Officials: Iqbal (Ike) Ahmed, MD, Study Director — Prism Eye Institute
Locations (5):
- United States (5):
  - Elios Vision Clinical Site, Glendale, Arizona
  - Elios Vision Clinical Site, Largo, Florida
  - Elios Vision Clinical Site, Rock Island, Illinois
  - Elios Vision Clinical Site, Oklahoma City, Oklahoma
  - Elios Vision Clinical Site, Kenosha, Wisconsin

IPD SHARING:
Plan to Share IPD: No